CLINICAL TRIAL: NCT02611700
Title: An Prospective, Multicenter, Double-blind, Randomized, Controlled Clinical Study of Nimotuzumab Combined With Paclitaxel and Cisplatin as First-line Treatment of Metastatic Esophageal Squamous Cell Carcinomas
Brief Title: Nimotuzumab in Combined With Paclitaxel and Cisplatin for Treatment of Metastatic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPL-IST-ESO-057
Record Dates: First submitted 2015-11-12; First posted 2015-11-23 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Esophageal Squamous Cell Carcinomas
MeSH Terms: interventions — nimotuzumab; Paclitaxel; Cisplatin; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): Nimotuzumab+TP(paclitaxel+cisplatin)
  Interventions: Drug: Nimotuzumab; Drug: Paclitaxel; Drug: Cisplatin
- control group (Placebo Comparator): Placebo + TP(paclitaxel+cisplatin)
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Placebo

INTERVENTIONS:
Drug: Nimotuzumab — 400mg,day1,weekly,until disease progression or toxicity
  Arms: experimental group
Drug: Paclitaxel — 175mg/m^2,for 3 hour(Peripherally Inserted Central Catheter,PICC),day1,21 days for a cycle ,until disease progression or toxicity，maximum duration is 6 cycles.
  Other Names: Paclitaxel Injection
Drug: Cisplatin — 60mg/m^2,day1，21 days for a cycle ,until disease progression or toxicity,maximum duration is 6 cycles.
  Other Names: Cisplatin for Injection
Drug: Placebo — 400mg,day1,weekly,until disease progression or toxicity
  Other Names: Nimotuzumab Placebo
  Arms: control group

SUMMARY:
This clinical study is designed as a phase 3,multicenter, double-blind, randomized, controlled study,to evaluate the efficacy and safety of nimotuzumab combined with paclitaxel+cisplatin（TP) compared with TP as first-line treatment for the metastatic esophageal squamous carcinoma.

DETAILED DESCRIPTION:
This clinical study is designed as a phase 3,multicenter, double-blind, randomized, controlled study,to evaluate the efficacy and safety of nimotuzumab combined with TP compared with TP as first-line treatment for the metastatic esophageal squamous carcinoma.The main endpoint is OS.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and sign a consent form;
2. Age≥18 years;
3. Histological diagnosis as metastatic esophageal squamous cell carcinoma, including: (1)Naked metastatic esophageal cancer：have no opportunity to receive any radical surgery or radical radiation therapy (2) recurrent metastatic esophageal cancer：recurrence after surgery or adjuvant radiotherapy or radical concurrent radio or radiochemotherapy,haven't received systemic chemotherapy and have measurable lesions outside radiotherapy target zone(3) recurrent metastatic esophageal cancer,more than 6 months after neoadjuvant or adjuvant chemotherapy;
4. When patients need to receive palliative radiotherapy,the palliative radiotherapy should complete over 4 weeks and target lesions should outside the radiotherapy target zone(radiotherapy lesions include but not limited to primary tumors, bone, lymph nodes);
5. According to RECIST 1.1 criteria, at least one measurable lesion exist;
6. Expected survival time is over 3 months;
7. Eastern Cooperative Oncology Group（ECOG）0 or 1;
8. Normal bone marrow and hematopoietic function;total bilirubin acuities≤1.5×Upper Limit Of Normal（ULN）, creatinine≤1.0×ULN, aspartate aminotransferase（AST）/alanine aminotransferase（ALT）≤2.5×ULN, ALP≤5.0×ULN, creatinine clearance > 60 ml/min, liver metastases patients: AST/ALT≤5.0×ULN;
9. Take effective contraceptive measures when in growth period;
10. Compliance is good.

Exclusion Criteria:

1. Have received any palliative chemotherapy for metastatic esophageal cancer
2. Recurrence or metastasis after neoadjuvant chemotherapy or postoperative adjuvant < 6 months;
3. Received any kinds of radiotherapy within 4 weeks;
4. Patients who can received palliative radiotherapy and all lesions are in one radiation zone;
5. Had received adjuvant/neoadjuvant therapy and have used paclitaxel within 6 months;
6. Had received adjuvant/neoadjuvant therapy and the cumulative dose of cisplatin was over 300 mg/m2;
7. Alone or combined with brain metastasis;
8. No measurable tumor lesions;
9. Combined with other primary malignant tumors (except cured skin basal cell carcinoma and cervical carcinoma in situ);
10. Allergy to the component of investigational drugs;
11. Patients who are receiving the treatment of chronic or multiple doses of corticosteroids (inhaled steroids or short-term oral cortisol according to the clinical indications were allowed);
12. Haven't recovered to degree 1 from the toxicity of treatment before.
13. Concomitant with severe cardiovascular diseases, such as uncontrol heart failure, coronary heart disease, cardiomyopathy, arrhythmia,high blood pressure or history of myocardial infarction within 5 years;
14. Concomitant with serious complications, such as the activity of the digestive tract hemorrhage, perforation, severe jaundice, gastrointestinal obstruction, active clinical infection (> 2 levels of infection standard);
15. With chronic diarrhea disease and renal insufficiency;
16. Have disease affecting cognition or mental abnormal;
17. Have other severe acute or chronic diseases;
18. Pregnancy or lactation women;
19. Have participated in other clinical trials within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Median time of overall survival(OS) | Up to 12 months
  Record all the survival status of each patient and calculate the median OS of all the patients

SECONDARY OUTCOMES:
Median time of progression-free survival（PFS） | Up to 12 months
  PFS is the time that passes from the date of signing Informed Consent Form（ICF）to the data on which "progresses" or the date on which the patient dies from any cause. The definition of "progression" since this generally involves imaging techniques(CT,MRI,et al).The Response Evaluation Criteria In Solid Tumors (RECISIT) 1.1 criteria will be used to evaluate "progression".The imaging evaluation will be done every 6 weeks.
Objective response rate（ORR） | Up to 12 months
  This wil be evaluated by RECISIT 1.1 criteria.It is dependent on imaging evaluation which will be done every 6 weeks. ORR is the percent of the patient who is evaluated as complete response(CR) or partial response (PR),that is (CR+PR)%.
Quality of life | baseline;once every 6 weeks until progression(6 weeks,12 weeks,18 weeks,up to 52 weeks)
  Using the European Organization for Research and Treatment of Cancer（EORTC）quality of life questionnaire（QLQ）-C30（Version3.0）and EORTC QLQ - OES18 to evaluate the quality of life of patients. The patients will fill this questionnaire when signing the ICF(as baseline) and every 6 weeks during treatment,until disease progression,up to 52 weeks. The progression is from date of randomization until the date of first documented progression or date of death from any cause.
Incidence of adverse events | Up to 30 days after last administration of nimotuzumab

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Dr, Study Chair — Peking University Cancer Hospital & Institute
Locations (27):
- China (27):
  - AnHui Provincial Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital Medical School of Chinese PLA, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The 307 Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center Sun Yat-Sen University Cancer Hospital, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - HuNan Cancer Hospital, Changsha, Hunan
  - JiangSu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital ,JiangNan University, Wuxi, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - LiaoNing Cancer Hospital, Shenyang, Liaoning
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Rui Jin Hospital Shanghai Jiao Tong University School Of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan hospital of fudan university, Shanghai, Shanghai Municipality
  - The First Affiliated of Xi'an Communication University, Xi’an, Shanxi
  - XiJing Hospital, Xi’an, Shanxi
  - West China Hospital,SiChuan University, Chengdu, Sichuan
  - TianJin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hostpital School of Medicine,Zhejiang University, Hangzhou, Zhejiang
  - The second Affiliated hospital of Zhejiang University School o, Hangzhou, Zhejiang
  - Zhejiang cancer hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided